CLINICAL TRIAL: NCT04704102
Title: Effects of Soft Tissue Mobilization of Neck Muscles in Individuals With Myogenous Temporomandibular Disorders: Muscle Energy Technique and Strain-counterstrain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University (Other)
Responsible Party: Principal Investigator, Lin Yang-Hua, Associate Professor, Chang Gung University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 2010280044
Record Dates: First submitted 2021-01-08; First posted 2021-01-11 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-07

CONDITIONS: Myogenous Temporomandibular Disorders (mTMD)
Keywords: myogenous temporomandibular disorders, neck pain, muscle energy technique, strain-counterstrain, head-neck posture
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Intervention Model Description: Include elements of both longitudinal (three groups) and cross-sectional (four-weeks intervention) research designs
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Muscle energy technique group (Experimental): Use one of the muscle energy technique methods -- postisometric relaxation technique(PIR) as the intervention method.
  Interventions: Behavioral: Muscle energy technique (MET)
- Strain-counterstrain group (Experimental): Use the Strain-counterstrain technique as the intervention method.
  Interventions: Behavioral: Strain-counterstrain (SCS)
- Control group (Sham Comparator): Use the modified Strain-counterstrain technique as the intervention method.
  Interventions: Behavioral: sham SCS

INTERVENTIONS:
Behavioral: Muscle energy technique (MET) — A manual therapy technique that uses the gentle muscle contractions of the patient to relax and lengthen muscles and normalize joint motion.
  Arms: Muscle energy technique group
Behavioral: Strain-counterstrain (SCS) — It's also called the "positional release technique", a manual therapy technique that passively positions the hypertonic (spasmed) muscles and dysfunctional joints in positions of shortened or comfort.
  Arms: Strain-counterstrain group
Behavioral: sham SCS — SCS intervention that position with opposite site limb and direction, and with modified method as consider the easiness of a practitioner to press the tender points
  Arms: Control group

SUMMARY:
This is a prospective case series study.There were 20 individuals with chronic neck pain accompanied by myogenous temporomandibular disorders(mTMD) from Linkou and Taoyuan Chang Gung hospitals, and Chang-Gung university. The purpose of this study was, first, to investigate the effects of muscle energy technique (MET) or strain-counterstrain (SCS) applied on the tender or trigger points of neck muscles on improving pain and pressure pain sensitivity in neck and masticatory muscles, the maximal mouth-opening range of motion, chewing endurance, and head-neck-shoulder posture in patients with chronic neck pain accompanied by mTMD. Second, whether the significant effects could be reached within the four-week intervention duration.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20~65
* Self-report neck pain ≥3 months (pain occurs between superior nuchal line and 1st level of thoracic spine)
* At least one tender point at both Upper trapezius and Sternocleidomastoid muscles
* Diagnosed as mTMD according to the Diagnostic Criteria for Temporomandibular Disorders(DC/TMD)

Exclusion Criteria:

* Cognitive deficit
* Malignancy, infection, cervical or orthognathic surgery, acute pain, and history of trauma in craniocervical region
* Neurological problem or cervical radiculopathy/myelopathy
* Cervical instability with positive rotational alar ligament stress test and transverse ligament stress test, jaw dislocation
* Tooth implantation or extraction a week before study
* Vertebrobasilar insufficiency

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Pain intensity in neck and masticatory muscles | 4 weeks
  ask participants the self-report pain intensity with the NPRS scale
Tenderness sensitivity in neck and masticatory muscles | 4 weeks
  measure the pressure pain threshold with digital pressure algometer

SECONDARY OUTCOMES:
Maximal mouth-opening | 4 weeks
  measure the maximal pain free mouth-opening distance
Chewing endurance | 4 weeks
  test for 5 minutes with chewing gum in the affected site
Head-neck-shoulder posture | 4 weeks
  measure the Head tilt angle(HTA), Craniovertebral angle(CVA) & Forward shoulder angle (FSA) by Photography in sagittal plane

CONTACTS AND LOCATIONS:
Locations (1):
- Yang-Hua, Lin, Taoyuan District, Taiwan